CLINICAL TRIAL: NCT03664934
Title: Pathophysiological Mechanism Behind Prolonged Whiplash Associated Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Anneli Peolsson, Professor, PhD, PT, Linkoeping University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Linköping University
Record Dates: First submitted 2018-08-28; First posted 2018-09-11 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Whiplash Injuries
Keywords: Neck pain, Rehabilitation, Muscles, Clinical Trial,; Diagnostics
MeSH Terms: conditions — Whiplash Injuries; Neck Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor blinded if a patient or a healthy control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients, Neck-specific exercises (Experimental): Patients before and after neck-specific exercises, subgroup to NCT01528579 with additional measures
  Interventions: Other: Exercises
- Healthy controls (No Intervention): Healthy controls, no treatment

INTERVENTIONS:
Other: Exercises — Neck-specific exercises for chronic whiplash associated disorders
  Other Names: No treatment, controls only
  Arms: Patients, Neck-specific exercises

SUMMARY:
The knowledge of pathophysiological mechanisms behind prolonged Whiplash Associated Disorders (WAD) is insufficient and whether changes can be restored by rehabilitation or not is unknown. The aim of these studies are to investigate different parameters to further learn about pathophysiological mechanisms (neck muscle fatty infiltration, cross-sectional area, volume, inflammation and function, brain structure and activity, biomarkers for stress and inflammation, cervical kinaesthesia and balance before and after intervention) and the association for clinical outcomes in individuals with chronic WAD (n=30) compared with age and gender matched healthy individuals (n=30). Measurements will be made at baseline (patients and healthy) and at 3 months (patients only, at the end of treatment). However, for the blood and saliva samples, they will be re-investigated in the healthy group as well. The study results may contribute to the development of improved understanding and diagnostics in chronic WAD that may improve future rehabilitation.

DETAILED DESCRIPTION:
BACKGROUND There is no consensus regarding the injury mechanism in complex prolonged Whiplash Associated Disorders (WAD) cases. Often, tissue damage and physiological alterations is not detectable. In order to improve future rehabilitation, a greater understanding of the mechanisms underlying whiplash injury and their importance for treatment success is required. It is also important to investigate if pathophysiological changes can be restored by rehabilitation.

AIM The projects aims to investigate neck muscle structure and function, biomarkers and the association with pain, disability and other outcomes before and after neck-specific exercises.

METHODS Design These are sub-group trials, each one independent of the others, in a prospective, multicentre, randomized controlled trial (RCT) with two parallel treatment arms conducted according to a protocol established before recruitment started (ClinicalTrials.gov Protocol ID: NCT03022812). Physiotherapist-led neck-specific exercise previously shown to be effective for the current population constitutes the control treatment for the new Internet-based neck-specific exercise treatment. In the RCT, a total of 140 patients will be included (70 from each group), whereof 30 (both randomization arms equally) consecutively will be asked to participate in the present sub-group study. The sub-group studies aims to start September 2019. Independent physiotherapists in primary health care will distribute the treatment.

In sub-group of individuals, additional measurements will be performed before and after interventions end (3 months follow-up). The physical measurements will be performed by independent specially trained test-leaders blinded to randomization.

Additionally, 30 neck healthy individuals without serious diseases matched for age and gender will consecutively be investigated.

Study population

The inclusion criteria for patients are:

* Chronic neck problems corresponding to WAD grades 2-3 verified by clinical examination
* Average estimated pain in the last week at least 20 mm on the visual analogue scale (VAS)
* Neck disability of more than 20% on the Neck Disability Index (NDI) [10]
* Working age (18 - 63 years)
* Daily access to a computer/tablet/smart phone and Internet
* Neck symptoms within the first week after the injury (i.e., neck pain, neck stiffness, or cervical radiculopathy).

For the present sub group study additional criteria were:

* Right handed
* Dominant right sided or equal sided pain

Inclusion criteria for healthy controls:

• Age and gender matched healthy individuals without neck pain and disability (VAS <10mm, NDI <5%) that feel overall healthy without known diseases.

Exclusion criteria for patients:

* Individuals with any of the following signs of head injury at the time of whiplash injury will be excluded: loss of consciousness, amnesia before or after the injury, altered mental status (e.g., confusion, disorientation), focal neurological changes (changes in smell and taste).
* Previous fractures or dislocation of the cervical spine
* Known or suspected serious physical pathology included myelopathy,
* Spinal tumours
* Spinal infection
* Ongoing malignancy
* Previous severe neck problems that resulted in sick leave for more than a month in the year before the current whiplash injury
* surgery in the cervical spine
* Generalized or more dominant pain elsewhere in the body
* Other illness/injury that may prevent full participation
* Inability to understand and write in Swedish

Additional criteria in the present sub group:

* Increased risk of bleeding,
* BMI >35
* Contraindications of MRI such as metal, severe obesity, pacemaker and pregnancy.

Exclusion criteria for healthy controls:

* Earlier neck injury,
* Recurrent neck pain,
* Earlier treatment for neck pain.
* Increased risk of bleeding,
* BMI >35
* Contraindications of MRI

Recruitment and randomization Information about the study will be provided by healthcare providers, reports in newspapers, social media, and the university's website. Interested patients will contact the research team through the project website. After completing a small survey on the website, a project team member (physiotherapist) will perform a telephone interview and ask about the patient's medical history. An appointment for a physical examination and additional interview for the present sub-group study is made as a last step to ensure that the criteria for study participation are met. If the study criteria are met, written and oral informed consent are obtained, and the patient will fill out a questionnaire and undergo physical measurements of neck-related function. Baseline measurements must be completed for inclusion.

Healthy individuals will consecutively be recruited among friends, family and staff at the university or the university hospital to suit the age and gender of a patient.

Intervention for the patient group The intervention consists of neck-specific exercises distributed in two different ways, twice a week at the physiotherapist clinic for 3 months (NSE group) or with 4 physiotherapy visits only combined with a web-based system (NSEIT group).

A. In the NSE group, patients will get an explanation and justification for the exercise consisting of basic information about the musculoskeletal anatomy of the neck relevant to the exercises given by the physiotherapist in order to motivate the patient and help make them feel safe and reassured. The patients undergo a 12-week training programme with a physiotherapist 2 days/week (total 24 times). Exercises are chosen from a clear and written frame of exercises. The training includes exercises for the deep neck muscles, continuing with the endurance training of neck and shoulder muscles. The exercises are individually adjusted according to the individual's physical conditions and progressively increased in severity and dose. Exercise-related pain provocation is not accepted. The patient may also perform exercises at home. At the end of the treatment period, the participants are encouraged to continue practising on their own. The exercises have been used with good results in previous RCTs.

B. In the NSEIT group, patients will receive the same information and training programmes as the NSE group, but with 4 visits to the physiotherapist instead of 24. Exercises are introduced, progressed, and followed up to ensure correct performance. The exercises are performed and most of the information is given with the help of Internet support outside the healthcare system. Photos and videos of the exercises (a clear stepwise progression) and information are available on the Web-based system. A SMS reminder is automatically available if the exercise diary is not completed. The time required for training is the same as in group A, but without the patient having to go to the physiotherapy clinic. The Internet programme was developed by experienced physiotherapists/ researchers together with technicians and clinicians. Technicians are available to assist the participants if any technical difficulties arise. The patients will be introduced to the exercises and get information and support at the physiotherapy visits.

Variables and measurements Background data and data in the RCT include personal details, questionnaires and test results regarding pain, physical and psychological functioning, health and cost-effectiveness described elsewhere (ClinicalTrials.gov Protocol ID: NCT03022812).

Measurements will be done at baseline for both groups and at 3 months follow-up for the patient when treatment ends. Except for blood and saliva samples that will be collected twice (baseline and repeated after 3 months), the measurements will be performed at baseline only for the healthy individuals.

ELIGIBILITY:
Study population

The inclusion criteria for patients are:

* Chronic neck problems corresponding to WAD grades 2-3 verified by clinical examination
* Average estimated pain in the last week at least 20 mm on the visual analogue scale (VAS)
* Neck disability of more than 20% on the Neck Disability Index (NDI) [10]
* Working age (18 - 63 years)
* Daily access to a computer/tablet/smart phone and Internet
* Neck symptoms within the first week after the injury (i.e., neck pain, neck stiffness, or cervical radiculopathy).

For the present sub group study additional criteria were:

* Right handed
* Dominant right sided or equal sided pain

Inclusion criteria for healthy controls:

• Age and gender matched healthy individuals without neck pain and disability (VAS <10mm, NDI <5%) that feel overall healthy without known diseases.

Exclusion criteria for patients:

* Individuals with any of the following signs of head injury at the time of whiplash injury will be excluded: loss of consciousness, amnesia before or after the injury, altered mental status (e.g., confusion, disorientation), focal neurological changes (changes in smell and taste).
* Previous fractures or dislocation of the cervical spine
* Known or suspected serious physical pathology included myelopathy,
* Spinal tumours
* Spinal infection
* Ongoing malignancy
* Previous severe neck problems that resulted in sick leave for more than a month in the year before the current whiplash injury
* surgery in the cervical spine
* Generalized or more dominant pain elsewhere in the body
* Other illness/injury that may prevent full participation
* Inability to understand and write in Swedish

Additional criteria in the present sub group:

* Increased risk of bleeding,
* BMI >35
* Contraindications of MRI such as metal, severe obesity, pacemaker and pregnancy.

Exclusion criteria for healthy controls:

* Earlier neck injury,
* Recurrent neck pain,
* Earlier treatment for neck pain.
* Increased risk of bleeding,
* BMI >35
* Contraindications of MRI such as metal, severe obesity, pacemaker and pregnancy.

Ages: 18 Years to 63 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2021-12-16 (Actual); Study Completion 2021-12-16 (Actual)

PRIMARY OUTCOMES:
Speckle tracking analyses of neck and shoulder muscle function | Baseline and at 3 months follow-up when intervention ended. The outcome measure is going to report a change over time for patients.
  Measured with medical ultrasonography during neck and arm exercises
Cross-sectional area, volume, fatty infiltration and inflammation of neck muscles | Baseline, 3 months. The outcome measure is going to report a change over time for patients.
  Neck and some whole body imaging measured with 3.0 T MRI scanner
Brain function in cortical networks related to pain | Baseline, 3 months. The outcome measure is going to report a change over time for patients.
  Measured with a resting-state fMRI protocol with an echo planar imaging (EPI) sequence
Biomarkers for inflammation and stress | Baseline, 3 months. The outcome measure is going to report a change over time for patients.
  Measured with blood samples and saliva
Cervikal kinaesthesia | Baseline, 3 months. The outcome measure is going to report a change over time for patients.
  Neck-eye coordination
Balance test | Baseline, 3 months. The outcome measure is going to report a change over time for patients.
  Postural sway during single and double leg stance

SECONDARY OUTCOMES:
Neck Disability Index (NDI) | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Self-reported neck-specific function. Score 0 to 50 (or in percentages 0% to 100%); 0p/0%=no disability, 50p/100%=complete activity limitation
Whiplash Disability Questionnaire | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Disability associated with whiplash, in patients. Score 0 to 130; 0=no disability, 130=maximum disability.
Patient-specific functional scale (PSFS) | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Individual ratings of function to quantify activity limitations, in patients. Score 0-10 score; 0= Unable to perform activity, 10= Able to perform activity at the same level as before injury or problem. Total score=sum of the activity scores/ number of activities.
Pain intensity in neck, head, and arm and dizziness by a Visual Analogue Scale (VAS) (0-100 mm; where 0=no pain, 100= worst imaginable pain ) | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Pain intensity. Score 0 to 100 mm; 0=no pain, 100=worst imaginable pain
Distribution of pain by a pain drawing assessed with images | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Distribution of pain, in patients
Frequency of pain | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Frequency of pain, in patients
Use of pain medications | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Use of pain medications, in patients
Dizziness/balance by the Dizziness Handicap Inventory (DHI) | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Dizziness questionnaire, in patients
Headache Questions by VAS and the Headache Impact Test (HIT-6) | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Impact of headache, in patients
Pain Catastrophizing Scale (PCS), total scores range from 0 - 52; 0=no catastrophizing, 52= maximum catastrophizing | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Self-reported pain catastrophizing, in patients
EuroQuol five dimensions | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Self-reported health, in patients
Effort Reward Imbalance questionnaire | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Work related balance between effort and reward, in patients
Symptoms Satisfaction scale | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Satisfaction with present symptoms, in patients. 1 to 7 scale; 1=delighted, 7=terrible.
Physical activity score, a combination score of the 2 questions (everyday physical activity and exercise/sport/open-air activity) to a combined 4-point score | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Physical activity. Score 0 to 4; 0=inactivity, 4=high activity.
Health care consumption, number of visits | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Health care consumption, in patients
Self-Efficacy Scale (SES) | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Self-reported self-efficacy, in patients. Score 0-200; 0=no self-efficacy, 200=strong self-efficacy
Fear Avoidance Beliefs Questionnaire (FABQ) | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Fear Avoidance Beliefs, in patients
Hospital Anxiety and Depression Scale (HAD) | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Depression and anxiety. Each subscale (depression and anxiety) range from 0 to 21; 0=normal, 21=severe
Post Traumatic Stress Disorder checklist (PCL-S) | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Post Traumatic Stress, in patients
Range of neck motion | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Range of motion, in patients
Ergonomics questions and how work is perceived | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Work ergonomics, in patients
Sickness presence by the Stanford presenteeism scale (SPS-6) | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Sickness presence at work, impact of health problems on individual work performance and overall perceived productivity , in patients. Scores 6-30, with lower scores indicting lower Presenteeism, and higher scores indicating higher Presenteeism.
Patient Enablement Instrument (PEI) questionnaire | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Patient enablement, in patients
Consumption of analgesic drugs prescribed through the drug registry | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Consumption of analgesic drugs, in patients
Sick-leave registration, number of days and episodes | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Sick-leave, in patients
Cognitive failures questionnaire (CFQ) | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Cognitive function, in patients
Sensorimotor control of the neck muscles, mm Hg | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Sensorimotor control, in patients
Neck muscle endurance of ventral and dorsal neck muscles in seconds | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Neck muscle endurance, in patients
Balance measured in seconds, standing on one leg with eyes closed | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Balance, in patients
Neurology | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Clinical examination of neurology, in patients, such as reflexes, sensibility, muscle weakness, Spurling´s test, neural tension test.
Work Ability Index (WAI) | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Self-reported work ability, in patients
Global rating of change scale | Change from baseline to 3 months (the end of treatment) and 15 months (1 year after study treatment is finalized) follow-up
  Overall change because of the treatment, in patients. Score -5 (very much worse to +5 completely recovered and importance of change 0=not at all important, 100= very important.

OTHER OUTCOMES:
Background data such as age and gender, living circumstances | Baseline
  Background data such as age, gender, living circumstances

CONTACTS AND LOCATIONS:
Overall Officials: Anneli Peolsson, Professor, Principal Investigator — Linkoeping University
Locations (1):
- Linköping University, Linköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Unidentified data may be available upon resonable request (may need approval from the ethics comittee as it contains data about health).

REFERENCES:
- [Derived] Ragnarsdottir H, Peterson G, Gislason MK, Oddsdottir GL, Peolsson A. The effect of a neck-specific exercise program on cervical kinesthesia for patients with chronic whiplash-associated disorders: a case-control study. BMC Musculoskelet Disord. 2024 May 2;25(1):346. doi: 10.1186/s12891-024-07427-9. PMID 38693515
- [Derived] Peolsson A, Karlsson A, Ghafouri B, Ebbers T, Engstrom M, Jonsson M, Wahlen K, Romu T, Borga M, Kristjansson E, Bahat HS, German D, Zsigmond P, Peterson G. Pathophysiology behind prolonged whiplash associated disorders: study protocol for an experimental study. BMC Musculoskelet Disord. 2019 Feb 2;20(1):51. doi: 10.1186/s12891-019-2433-3. PMID 30711003

DOCUMENTS (3):
  • Study Protocol (2018-08-31): https://cdn.clinicaltrials.gov/large-docs/34/NCT03664934/Prot_001.pdf
  • Statistical Analysis Plan (2018-08-31): https://cdn.clinicaltrials.gov/large-docs/34/NCT03664934/SAP_000.pdf
  • Informed Consent Form (2018-09-06): https://cdn.clinicaltrials.gov/large-docs/34/NCT03664934/ICF_002.pdf